CLINICAL TRIAL: NCT04487860
Title: A Phase II, Randomized, Double Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Efficacy and Safety of AS012 in Subjects With Non-segmental Vitiligo
Brief Title: Efficacy and Safety of AS012 in Subjects With Non-segmental Vitiligo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AS012-20-01
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Results first posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2022-06

CONDITIONS: Non-segmental Vitiligo

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- AS012 dose regimen I (Experimental): Oral
  Interventions: Drug: AS012
- AS012 dose regimen II (Experimental): Oral
  Interventions: Drug: AS012
- AS012 dose regimen III (Experimental): Oral
  Interventions: Drug: AS012
- AS012 dose regimen IV (Experimental): Oral
  Interventions: Drug: AS012
- Placebo (Placebo Comparator): Oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AS012 — oral administration
  Arms: AS012 dose regimen I; AS012 dose regimen II; AS012 dose regimen III; AS012 dose regimen IV
Drug: Placebo — oral administration
  Arms: Placebo

SUMMARY:
This is a randomized, double blind, placebo-controlled, phase II study. The study will be performed as a multicenter, multinational study.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent.
2. Male or female ≥ 18 years of age at time of screening
3. Stable (without new patches ≥ 1 year) or unstable (with new patches for the last 1 year) vitiligo
4. VASI of ≥ 4 at screening and baseline

Exclusion Criteria:

1. Segmental vitiligo, focal, or mixed Vitiligo
2. Subjects who have high risk of suicidality at the Screening assessment based on Investigator's judgment
3. History of alcohol or drug abuse in the previous 2 years
4. Subjects who were submitted to melanocyte transfer

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2023-02-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- United States (19):
  - Sun Pharma Site 15, Phoenix, Arizona
  - Sun Pharma Site 02, Bryant, Arkansas
  - Sun Pharma Site 09, Fremont, California
  - Sun pharma site 30, Los Angeles, California
  - Sun Pharma Site 01, Brandon, Florida
  - Sun Pharma Site 06, Fort Lauderdale, Florida
  - Sun Pharma Site 04, Miami, Florida
  - Sun Pharma Site 05, Miramar, Florida
  - Sun Pharma Site 10, Ormond Beach, Florida
  - Sun Pharma Site 14, West Lafayette, Indiana
  - Sun Pharma Site 12, Baton Rouge, Louisiana
  - Sun Pharma Site 13, New Orleans, Louisiana
  - Sun pharma site 31, Boston, Massachusetts
  - Sun Pharma Site 07, Troy, Michigan
  - Sun Pharma Site 29, East Greenwich, Rhode Island
  - Sun Pharma Site 08, Warwick, Rhode Island
  - Sun Pharma Site 03, Dallas, Texas
  - Sun Pharma Site 16, Pflugerville, Texas
  - Sun Pharma Site 11, Mill Creek, Washington
- India (12):
  - Sun Pharma Site 19, Ahmedabad, Gujarat
  - Sun Pharma Site 20, Gandhinagar, Gujarat
  - Sun Pharma Site 28, Rajkot, Gujarat
  - Sun Pharma Site 23, Bangalore, Karnataka
  - Sun PharmaSite 24, Mysuru, Karnataka
  - Sun Pharma Site 21, Aurangabad, Maharashtra
  - Sun Pharma Site 25, Nashik, Maharashtra
  - Sun Pharma Site 26, Pune, Maharashtra
  - Sun Pharma Site 17, Rājsamand, Rajasthan
  - Sun Pharma Site 27, Lucknow, Uttar Pradesh
  - Sun Pharma Site 18, Lucknow, Uttar Pradesh
  - Sun Pharma Site 22, Chandigarh

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Part I: Up to 24 weeks: Subjects were randomized to Placebo
  Part II: week 24 to week 52: No Subjects
  Part III: week 52 to week 64: No Subjects
- Placebo to AS012 Dose Regimen II at Week 24: Part I: Up to 24 weeks: No subjects
  Part II: week 24 to week 52: Subjects initially randomized to placebo were rerandomized to AS012 dose 2x
  Part III: week 52 to week 64: After week 52, the study treatment was stopped and all subjects entered the follow-up period to monitor safety and tolerability for 12 weeks after the last dose of study treatment.
- Placebo to AS012 Dose Regimen IV at Week 24: Part I: Up to 24 weeks: No subjects
  Part II: week 24 to week 52: Subjects initially randomized to placebo were rerandomized to AS012 dose 6x
  Part III: week 52 to week 64: After week 52, the study treatment was stopped and all subjects entered the follow-up period to monitor safety and tolerability for 12 weeks after the last dose of study treatment.
- AS012 Dose Regimen I: Part I: Up to 24 weeks: Subjects were randomized to AS012 dose x
  Part II: week 24 to week 52: Subjects originally randomized to AS012 doses remained on their assigned dosing regimen until the end of Part II (week 52).
  Part III: week 52 to week 64: After week 52,the study treatment was stopped and all subjects entered the follow-up period to monitor safety and tolerability for 12 weeks after the last dose of study treatment.
- AS012 Dose Regimen II: Part I: Up to 24 weeks: Subjects were randomized to AS012 dose 2x
  Part II: week 24 to week 52: Subjects originally randomized to AS012 doses remained on their assigned dosing regimen until the end of Part II (week 52).
  Part III: week 52 to week 64: After week 52, the study treatment was stopped and all subjects entered the follow-up period to monitor safety and tolerability for 12 weeks after the last dose of study treatment.
- AS012 Dose Regimen III: Part I: Up to 24 weeks: Subjects were randomized to AS012 dose 4x
  Part II: week 24 to week 52: Subjects originally randomized to AS012 doses remained on their assigned dosing regimen until the end of Part II (week 52).
  Part III: week 52 to week 64: After week 52, the study treatment was stopped and all subjects entered the follow-up period to monitor safety and tolerability for 12 weeks after the last dose of study treatment.
- AS012 Dose Regimen IV: Part I: Up to 24 weeks: Subjects were randomized to AS012 dose 6x
  Part II: week 24 to week 52: Subjects originally randomized to AS012 doses remained on their assigned dosing regimen until the end of Part II (week 52).
  Part III: week 52 to week 64: After week 52 the study treatment was stopped and all subjects entered the follow-up period to monitor safety and tolerability for 12 weeks after the last dose of study treatment.
Period: Part 1
Arm/Group | Placebo | Placebo to AS012 Dose Regimen II at Week 24 | Placebo to AS012 Dose Regimen IV at Week 24 | AS012 Dose Regimen I | AS012 Dose Regimen II | AS012 Dose Regimen III | AS012 Dose Regimen IV
Started | 59 | 0 | 0 | 62 | 71 | 63 | 72
Completed | 40 | 0 | 0 | 44 | 59 | 46 | 54
Not Completed | 19 | 0 | 0 | 18 | 12 | 17 | 18
Period: Part 2
Arm/Group | Placebo | Placebo to AS012 Dose Regimen II at Week 24 | Placebo to AS012 Dose Regimen IV at Week 24 | AS012 Dose Regimen I | AS012 Dose Regimen II | AS012 Dose Regimen III | AS012 Dose Regimen IV
Started | 0 | 20 | 20 | 44 | 59 | 46 | 54
Completed | 0 | 12 | 14 | 28 | 36 | 34 | 38
Not Completed | 0 | 8 | 6 | 16 | 23 | 12 | 16
Period: Part 3
Arm/Group | Placebo | Placebo to AS012 Dose Regimen II at Week 24 | Placebo to AS012 Dose Regimen IV at Week 24 | AS012 Dose Regimen I | AS012 Dose Regimen II | AS012 Dose Regimen III | AS012 Dose Regimen IV
Started | 0 | 12 | 14 | 28 | 36 | 34 | 38
Completed | 0 | 11 | 14 | 27 | 35 | 31 | 34
Not Completed | 0 | 1 | 0 | 1 | 1 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo
- Placebo to AS012 Dose Regimen II at Week 24: Placebo to AS012 dose 2x at Week 24
- Placebo to AS012 Dose Regimen IV at Week 24: Placebo to AS012 dose 6x at Week 24
- AS012 Dose Regimen I: AS012 dose x
- AS012 Dose Regimen II: AS012 dose 2x
- AS012 Dose Regimen III: AS012 dose 4x
- AS012 Dose Regimen IV: AS012 dose 6x
- Total: Total of all reporting groups
Arm/Group | Placebo | Placebo to AS012 Dose Regimen II at Week 24 | Placebo to AS012 Dose Regimen IV at Week 24 | AS012 Dose Regimen I | AS012 Dose Regimen II | AS012 Dose Regimen III | AS012 Dose Regimen IV | Total
Number analyzed (Participants) | 59 | 20 | 20 | 62 | 71 | 63 | 72 | 367
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Subjects initially randomized to placebo were rerandomized to AS012 dose 2x or AS012 dose 6x in Part II of the study and therefore the data are reported separately for the "Placebo to AS012 Dose Regimen" arms.
  years
    Placebo and AS012 Regimens: number analyzed (Participants) | 59 | 0 | 0 | 62 | 71 | 63 | 72 | 327
    Placebo and AS012 Regimens | 44.2 (14.65) |  |  | 48.1 (14.85) | 45.2 (12.87) | 46.8 (14.52) | 41.8 (15.18) | 45.1 (14.49)
    Placebo to AS012 Regimens: number analyzed (Participants) | 0 | 20 | 20 | 0 | 0 | 0 | 0 | 40
    Placebo to AS012 Regimens |  | 45.6 (14.81) | 43.3 (16.76) |  |  |  |  | 44.5 (15.66)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Subjects initially randomized to placebo were rerandomized to AS012 dose 2x or AS012 dose 6x in Part II of the study and therefore the data are reported separately for the "Placebo to AS012 Dose Regimen" arms.
  Participants
    Placebo and AS012 Regimens: number analyzed (Participants) | 59 | 0 | 0 | 62 | 71 | 63 | 72 | 327
    Placebo and AS012 Regimens: Female | 31 | 0 | 0 | 32 | 38 | 36 | 34 | 171
    Placebo and AS012 Regimens: Male | 28 | 0 | 0 | 30 | 33 | 27 | 38 | 156
    Placebo to AS012 Regimens: number analyzed (Participants) | 0 | 20 | 20 | 0 | 0 | 0 | 0 | 40
    Placebo to AS012 Regimens: Female | 0 | 11 | 8 | 0 | 0 | 0 | 0 | 19
    Placebo to AS012 Regimens: Male | 0 | 9 | 12 | 0 | 0 | 0 | 0 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Subjects initially randomized to placebo were rerandomized to AS012 dose 2x or AS012 dose 6x in Part II of the study and therefore the data are reported separately for the "Placebo to AS012 Dose Regimen" arms.
  Participants
    Placebo and AS012 Regimens: number analyzed (Participants) | 59 | 0 | 0 | 62 | 71 | 63 | 72 | 327
    Placebo and AS012 Regimens: Hispanic or Latino | 19 | 0 | 0 | 18 | 17 | 15 | 16 | 85
    Placebo and AS012 Regimens: Not Hispanic or Latino | 40 | 0 | 0 | 44 | 54 | 48 | 56 | 242
    Placebo and AS012 Regimens: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Placebo to AS012 Regimens: number analyzed (Participants) | 0 | 20 | 20 | 0 | 0 | 0 | 0 | 40
    Placebo to AS012 Regimens: Hispanic or Latino | 0 | 8 | 6 | 0 | 0 | 0 | 0 | 14
    Placebo to AS012 Regimens: Not Hispanic or Latino | 0 | 12 | 14 | 0 | 0 | 0 | 0 | 26
    Placebo to AS012 Regimens: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Vitiligo Area Scoring Index Score
Description: Vitiligo Area Scoring Index score: numeric score that can range from 0 to 100, with higher VASI scores denoting poorer the disease state
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AS012 Dose Regimen I | AS012 Dose Regimen II | AS012 Dose Regimen III | AS012 Dose Regimen IV
Number analyzed (Participants) | 59 | 62 | 71 | 63 | 72
score on a scale | -0.472 (1.0422) | -0.271 (2.5139) | -0.706 (1.7301) | -1.145 (2.7721) | -0.110 (2.6168)
Statistical Analysis 1: Comparison: Placebo vs AS012 Dose Regimen I; Test type: Superiority; p = 0.7905, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs AS012 Dose Regimen II; Test type: Superiority; p = 0.7372, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs AS012 Dose Regimen III; Test type: Superiority; p = 0.2989, ANCOVA
Statistical Analysis 4: Comparison: Placebo vs AS012 Dose Regimen IV; Test type: Superiority; p = 0.3328, ANCOVA

2. Secondary Outcome: Mean Change From Baseline in Vitiligo Extent Score (VES) on Clinical Pictures
Description: The Vitiligo Extent Score (VES) measures the overall vitiligo involvement in the body based on clinical pictures reflecting the natural distribution of the disease across 19 body areas (e.g., face, trunk, arms, legs, hands, axillae, back, gluteal). For each area, one representative image is selected, assigning one of six degrees of involvement (1%, 5%, 10%, 25%, 50%, 75%). The total and final score is the sum of the measurements from all areas, calculated using a conversion table available in the online calculator (www.vitiligo-calculator.com), and expressed as the extension of body surface area affected (0-100). Higher scores indicate worse clinical involvement. The VES change from baseline to Week 24 was assessed for the ITT population.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AS012 Dose Regimen I | AS012 Dose Regimen II | AS012 Dose Regimen III | AS012 Dose Regimen IV
Number analyzed (Participants) | 59 | 62 | 71 | 63 | 72
score on a scale | -0.507 (1.7427) | -0.671 (2.2065) | -0.284 (2.4793) | -0.454 (2.1214) | -1.218 (3.3963)
Statistical Analysis 1: Comparison: Placebo vs AS012 Dose Regimen I; Test type: Superiority; p = 0.8989, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs AS012 Dose Regimen II; Test type: Superiority; p = 0.6768, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs AS012 Dose Regimen III; Test type: Superiority; p = 0.8209, ANCOVA
Statistical Analysis 4: Comparison: Placebo vs AS012 Dose Regimen IV; Test type: Superiority; p = 0.3106, ANCOVA

3. Secondary Outcome: Mean Change in Vitiligo Impact Patient Scale
Description: Subjects will be asked to complete a questionnaire to assess the burden experienced by individuals affected. For each of the statements in the Vitiligo Impact Patient Scale, 7 responses are suggested: always, very often, often, sometimes, rarely, never and not applicable. The individual answered as spontaneously as possible while thinking about their situation over the last 7 days. Summary scores range from 0 to 100. Higher values indicate a worse clinical condition.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AS012 Dose Regimen I | AS012 Dose Regimen II | AS012 Dose Regimen III | AS012 Dose Regimen IV
Number analyzed (Participants) | 59 | 62 | 71 | 63 | 72
score on a scale | -2.72 (12.575) | -3.48 (13.603) | -4.24 (18.984) | -2.50 (11.506) | -2.06 (15.082)
Statistical Analysis 1: Comparison: Placebo vs AS012 Dose Regimen I; Test type: Superiority; p = 0.8593, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs AS012 Dose Regimen II; Test type: Superiority; p = 0.9594, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs AS012 Dose Regimen III; Test type: Superiority; p = 0.9041, ANCOVA
Statistical Analysis 4: Comparison: Placebo vs AS012 Dose Regimen IV; Test type: Superiority; p = 0.7147, ANCOVA

4. Secondary Outcome: Physician's Global Assessment Scores
Description: Description: The investigator will perform an average assessment of all vitiligo lesions. The following scale will be used for the PGA: Score 0= No involvement, Score 1= Limited, Score 2= moderate, Score 3= Extensive or Score 4= Very extensive. Higher values indicate a worse clinical condition. The static Physician's Global Assessment determines vitiligo extend at a single point in time, without taking the baseline disease condition into consideration, in other words, represents the Proportion of subjects achieving a PGA score of "no involvement" (score 0) or "limited extent" (score 1) with at least 2-point reduction from Baseline Week 52.
Time Frame: Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo to AS012 Dose Regimen II at Week 24 | Placebo to AS012 Dose Regimen IV at Week 24 | AS012 Dose Regimen I | AS012 Dose Regimen II | AS012 Dose Regimen III | AS012 Dose Regimen IV
Number analyzed (Participants) | 12 | 14 | 27 | 36 | 34 | 38
Participants | 0 | 0 | 0 | 0 | 1 | 0

5. Secondary Outcome: Mean Change From Baseline in Dermatology Life Quality Index
Description: The DLQI scores are based on the response from the patient. Each question is scored from 0 (not affected at all) to 3 (very much affected). The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired OR lower scores indicate better quality of life.
Time Frame: Week 52
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo to AS012 Dose Regimen II at Week 24 | Placebo to AS012 Dose Regimen IV at Week 24 | AS012 Dose Regimen I | AS012 Dose Regimen II | AS012 Dose Regimen III | AS012 Dose Regimen IV
Number analyzed (Participants) | 12 | 14 | 28 | 36 | 34 | 38
score on a scale | 0.2 (2.12) | 0.0 (3.33) | -0.8 (3.08) | -0.6 (4.76) | -2.0 (3.49) | -0.2 (2.51)

ADVERSE EVENTS:
Time Frame: 64 Week
Description: The Safety Population will consist of all subjects who were randomized into the study and dispensed study drug. This population will be the primary population for the safety analysis.
  Subjects will be analyzed according to the actual treatment received
Groups:
- Placebo - Part I: Placebo - Part I
- AS012 Dose Regimen I- Part I: AS012 dose x- Part I
- AS012 Dose Regimen II - Part I: AS012 dose 2x- Part I
- AS012 Dose Regimen III - Part I: AS012 dose 4x- Part I
- AS012 Dose Regimen IV - Part I: AS012 dose 6x- Part I
- Placebo to AS012 Dose Regimen II at Week 24 - Part II: Placebo to AS012 dose 2x at Week 24 - Part II
- Placebo to AS012 Dose Regimen IV at Week 24 - Part II: Placebo to AS012 dose 6x at Week 24 - Part II
- AS012 Dose - Regimen I - Part II: AS012 dose X- Part II
- AS012 Dose Regimen II - Part II: AS012 dose 2 x - Part II
- AS012 Dose Regimen III - Part II: AS012 dose 4 x - Part II
- AS012 Dose Regimen IV - Part II: AS012 dose 6 x - Part II
- AS012 - Part III: treatment free
Arm/Group | Placebo - Part I | AS012 Dose Regimen I- Part I | AS012 Dose Regimen II - Part I | AS012 Dose Regimen III - Part I | AS012 Dose Regimen IV - Part I | Placebo to AS012 Dose Regimen II at Week 24 - Part II | Placebo to AS012 Dose Regimen IV at Week 24 - Part II | AS012 Dose - Regimen I - Part II | AS012 Dose Regimen II - Part II | AS012 Dose Regimen III - Part II | AS012 Dose Regimen IV - Part II | AS012 - Part III
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/62 | 0/70 | 0/63 | 0/72 | 0/20 | 0/20 | 0/44 | 0/59 | 0/46 | 0/54 | 0/162
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/62 | 0/70 | 0/63 | 0/72 | 0/20 | 0/20 | 0/44 | 0/59 | 0/46 | 0/54 | 0/162
Other Adverse Events (participants affected / at risk) | 0/59 | 0/62 | 0/70 | 0/63 | 0/72 | 1/20 | 0/20 | 0/44 | 0/59 | 0/46 | 0/54 | 0/162
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Part I (N=59) | AS012 Dose Regimen I- Part I (N=62) | AS012 Dose Regimen II - Part I (N=70) | AS012 Dose Regimen III - Part I (N=63) | AS012 Dose Regimen IV - Part I (N=72) | Placebo to AS012 Dose Regimen II at Week 24 - Part II (N=20) | Placebo to AS012 Dose Regimen IV at Week 24 - Part II (N=20) | AS012 Dose - Regimen I - Part II (N=44) | AS012 Dose Regimen II - Part II (N=59) | AS012 Dose Regimen III - Part II (N=46) | AS012 Dose Regimen IV - Part II (N=54) | AS012 - Part III (N=162)
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT04487860/Prot_002.pdf
  • Statistical Analysis Plan (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/60/NCT04487860/SAP_003.pdf